CLINICAL TRIAL: NCT05166447
Title: Twenty-year Follow-up of the Inter99 Cohort
Status: Enrolling by invitation | Type: Observational
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Steno Diabetes Center Copenhagen (Other); The Novo Nordisk Foundation Center for Basic Metabolic Research (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Allan Linneberg, Director, Professor, MD, PhD, Bispebjerg Hospital
Other Study IDs: INTER99 twenty year follow-up
Record Dates: First submitted 2021-08-26; First posted 2021-12-22 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Coronary Heart Disease; Acute Myocardial Infarction; Cardiovascular Diseases; Type 2 Diabetes; Obesity; Birth Weight
Keywords: type 2 diabetes; cardiovascular disease; fetal programming; birth weight; developmental origins of health and disease; obesity
MeSH Terms: conditions — Coronary Disease; Cardiovascular Diseases; Diabetes Mellitus, Type 2; Obesity; Birth Weight; Developmental Origins of Health and Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urine used in this project will be analyzed immediately and then destroyed. Participants will be asked for permission to store blood and urine in a biobank for future unspecified research that is not part of current project. The biological material will be stored in a biobank at the Center for Clinical Research and Prevention, Rigshospitalet, Glostrup, Denmark and/or at Steno Diabetes Center Copenhagen, Gentofte, Denmark. If participants grant permission, the material will be stored for 50 years or as long as national law allows. Biological material can only be used in a new research project with permission from the Regional Committee on Health Research Ethics Denmark for the Capital Region.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Being born small increases your risk of developing Type 2 diabetes (T2D) with age. Furthermore, data even suggest that some of the diseases ("complications") in the eyes, kidneys, nerves, liver, blood vessels and heart often seen in T2D patients may not only be due to high blood sugar levels, but rather they to some extent are due to reduced growth in your mother´s womb. The Inter99 cohort included 6784 Danish citizens aged 30 to 60 years when established 20 years ago. Data from the Inter99 cohort showed a strong role of low birth weight (LBW) on T2D risk. The aim is now to reexamine risk of T2D and complications in all the alive 6004 elderly Inter99 participants. Importantly, today there are available techniques to perform detailed examinations for even the earliest signs of complications in both subjects with and without diabetes, and the results of this study will altogether provide important new insights into both the origin and classification of T2D and associated complications. It is hypothesized that being born with lower birth weights increases the adult risk of T2D and heart disease and associated complications in the large and smaller blood vessels.

DETAILED DESCRIPTION:
BACKGROUND Type 2 Diabetes (T2D) affecting globally more than 400 million people represents one of the most significant global health challenges of our time. However, despite huge research investments, there are still limited insights into its complicated etiology and pathophysiology during the life-course. T2D is furthermore defined by arbitrary glycemic thresholds, which inadequately captures the diversity of clinical presentations and sub-phenotypes with differential complications and damages in multiple organs including small and large vessels, heart, kidney, liver and nerve tissue, often present already at the time of disease onset.

The heterogeneity of phenotypes in T2D is likely rooted in differential genetic, prenatal, and postnatal non-genetic etiologies between individuals. As for genetics, the known 568 T2D susceptibility variants are estimated to account for 18% of the putative genetic contribution to T2D. The totality of data from human famine catastrophes conclusively confirm the initial reports from Hertfordshire, UK, of an adverse intrauterine environment associated with low birth weight (LBW) playing a significant role in the development of T2D. The concept of fetal and early life developmental programming has been confirmed, validated and mechanistically examined in multiple animal studies. Studies in humans and animals have provided compelling evidence of an adverse fetal environment contributing to virtually all the known multiple organ defects influencing glucose homeostasis. Furthermore, emerging evidence consistently suggest that LBW and an adverse fetal environment play a direct and independent role in the development of important complications in T2D including cardiovascular disease, hypertension, dyslipidemia and vascular dysfunctions. Vascular stiffness reflected by elevated pulse-wave-velocity are early signs of micro- and/or macrovascular disease in patients with and without T2D. The fact that T2D patients often have a significant burden of vascular and metabolic complications already at diagnosis, indicates that factors influencing risk of T2D at the same time represent direct causes of co-morbidities that it is otherwise considered as complications to hyperglycemia. Accordingly, a distinct subgroup of T2D patients, as a result of an adverse fetal environment, may be affected by diabetic complications to a larger extent than patients with T2D due to other factors. Indeed, it was reported that LBW accounts for most of the excess cardiovascular disease (CVD) mortality in T2D. Moreover, LBW is associated with smaller kidneys with fewer nephrons and increased risk of chronic kidney disease. Another study reported increased risk of cardiac autonomic function (heart rate variability) in children, which is a known risk factor of CVD morbidity and mortality. Patients with T2D are at increased risk of developing NAFLD, which may progress to non-alcoholic stereo hepatitis (NASH), overt liver cirrhosis and liver cancer. NAFLD and NASH are clinically silent and under-diagnosed diseases with a global prevalence of 25-30% and is associated with increased risk of CVD in a non-genetic manner. Recent unpublished data from our group showed a threefold increased liver fat content in young, non-diabetic LBW men when studied before and after 4 weeks of a high carbohydrate challenge diet.

AIM To give a detailed phenotypical cardiometabolic description of the population-based Inter99-cohort, in order to examine associations of size at birth and prematurity, as proxies for the early fetal environment, concurrent lifestyle factors and genetic risk with the age-specific incidence of T2D and CVD, and its complications and co-morbidities, among Danish citizens aged 50-80 years.

HYPOTHESIS

1. An adverse fetal environment (LBW and/or prematurity) is associated with increased risk of developing a more severe T2D sub-phenotype with increased morbidity and mortality from micro- and macro vascular complications as well as cardiometabolic co-morbidities including NAFLD, compared with T2D patients born at term with a normal birth weight.
2. An adverse fetal environment is associated with increased morbidity and mortality from a range of micro- and macrovascular manifestations, as well as NAFLD, typically referred to as diabetes complications, even among elderly non- diabetic people with or without prediabetes (impaired glucose tolerance or impaired fasting glucose).

METHODS

The Inter99 study:

The population based Inter99 study was initiated in 1999 as a collaboration between Steno Diabetes Center Copenhagen (SDCC) and the Center for Clinical Research and Prevention (CCRP). From a population-based random sample of 61,301 30-60-year-old individuals living in the Western part of Copenhagen, Denmark, 13,016 people was invited to a health examination. The remaining control group (n=47,987) was followed in registries. The cohort was after baseline examination of 6,784 participants (52,5% acceptance rate), established as a randomized, non- pharmacological, lifestyle-counseling intervention study for prevention of diabetes and ischemic heart disease.

Clinical follow-up examinations after 5 years including glucose tolerance status had a participation rate of 66%, and the 10 years follow-up was based on registry data. While the lifestyle intervention had no effects on 5- or 10-year incidence rates of diabetes or cardiovascular disease, the in-depth clinical examinations of the cohort have contributed substantially to our knowledge of the etiology of T2D and associated traits. Original midwife records have been collected from 4.744 participants. Despite the relatively low average age of the cohort of only 46 years in 1999, a strong inverse relationship between birth weight and risk of T2D in this contemporary Danish population was confirmed. The prevalence of T2D associated retinal changes in the Inter99 cohort was studied in a subgroup of 970 participants. Interestingly, diabetic retinopathy was present in 7,5% of the 490 subjects with completely normal glucose tolerance, supporting the notion that factors other than elevated glucose contributes to the risk of diabetic complications.

Data collection:

The planned register-based study will include morbidity and mortality data from the newly established Danish Diabetes Register at SDCC. Biochemical data to estimate clinical trajectories following T2D diagnosis will be obtained from the Danish Clinical Laboratory Information System Research Database). Information on cardiovascular outcomes is based on the Danish National Patient Register. CVD is defined as ischaemic heart disease, heart failure, atherosclerotic macro-vascular disease, hypertensive disease, atrial fibrillation and cerebrovascular disease.

The 20-year cardiometabolic outcome follow-up study will include clinical examinations tailored to capture and expand our growing understanding of T2D subgroups, and with increased focus on T2D associated vascular and cardiometabolic co-morbidities and complications. The totality of data already available in the Inter99 cohort range from prenatal health information on birth weights and prematurity, glucose tolerance at baseline and 5 years follow-up, lifestyle and general health information including comprehensive Food Frequency Questionnaire data, numerous biomarkers and unparalleled genetic (GWAS) data. When subsequently combined with detailed Danish registries and our innovative clinical cardiometabolic deep phenotyping follow-up study, the cohort will constitute a hitherto unparalleled research platform to delineate the role of the fetal environment, as well as lifestyle and genetic determinants, for the development of T2D, its co-morbidities, as well as its clinical sub-phenotypes.

Examinations:

All individuals will be invited for a clinical examination at CCRP, Rigshospitalet, Glostrup, including:

1. Fasting blood samples for analysis of glucose, insulin, C-peptide, lipids, HbA1c, electrolytes, e-GFR, liver function test, extra plasma and serum for micronutrient status, metabolomics, lipidomics, transcriptomics, DNA and GAD-antibodies.
2. Urine for albumin, metabolomic and proteomic profiling.
3. Anthropometrics and body composition (bioelectrical impedance)
4. Liver stiffness by transient elastography (TE) will be used for noninvasive diagnosis of fibrosis and cirrhosis (FibroScan 502 Touch; Echosens, France).
5. Arterial stiffness and central (carotis-femoralis) pulse wave velocity (cfPWV) using the gold standard SphygmoCor© Pulse Wave method (AtCor Medical, Sydney, Australia).
6. Retinal fundus photo and optical coherence tomography (OCT) will be taken of both eyes with the Optos Ultra Widefield apparatus (Optos Monaco, Optos PLC, Dunfermline, UK) and images graded according to a modified version of the 'Proposed International Clinical DR severity scale' applying a deep learning (DL) algorithm by convolutional neural networks.
7. As a measure of cardiac autonomic neuropathy, simple bedside tests using heart rate variability (HRV) indices or response in heart rate to standing, slow breathing, or the Valsalva maneuver (cardiovascular autonomic reflex tests [CARTs]) will be used with a Vagus device (Medicus Engineering, Aarhus, Denmark).
8. Measurement of the electrical conduction system of the heart by ECG (electrocardiogram), using 12 electrodes.
9. Spirometry to measure pulmonary function i.e. expiratory forced vital capacity (FVC) and forced expiratory volume in one second (FEV1).
10. Handgrip strength will be used to measure maximum hand muscle strength. Handgrip strength is a strong predictor of both morbidity and mortality in the older population.
11. A 30 second sit to stand test will examine physical performance of participants, according to the number of times participants get to a full stand in 30 seconds.
12. Blood pressure (systolic and diastolic) is measured thrice with an electronic blood pressure monitor and fitting cuff after five minutes rest in sitting position.
13. Oxygen saturation will be measured

Participants will be asked to fill in validated questionnaires on general health, occurrence of chronic diseases, lifestyle factors and dietary intake.

On a separate occasion, participants will be invited for a coronary artery CT- calcium-scan (CCTA) at Dept. of Cardiology, Rigshospitalet (RH). CT-angiography will provide data on structural heart disease, coronary artery calcium score as well as subclinical obstructive coronary atherosclerosis, which all are associated with adverse long-term outcome. CT imaging will be performed using a 320- multidetector scanner (Aquilion One, Toshiba Medical Systems, Japan). A cardio- selective beta-blocker (metoprolol 25-150 mg) can be administered orally 1 h before scanning in participants with a heart rate of 60 bpm and no contraindications. Intravenous contrast media (Visipaque) will be used. A fixed- target protocol using one rotation acquisition with a prospective exposure window fixed at 350 ms centered at the 75% phase of the RR cycle will be used to restrict radiation dose.

A subset of participants will be asked:

* To wear a continuous glucose monitoring system (CGM) for two weeks to provide information about variability in glucose levels.
* To wear a physical activity monitor by Axivity to objectively measure physical activity and sedentary behavior by continuous 24-hour*7 days measurement using Axivity® AX3 accelerometers (www.axivity.com) skin-taped to the thigh.
* To participate in a dietary assessment study using a web-based dietary assessment software for seven consecutive days. The dietary assessment software is structured according to a typical Danish meal pattern covering breakfast, lunch, dinner and three in-between meals (morning, afternoon and evening).
* To participate in a 24-hour urine collection to estimate sodium and potassium intake using 24-hour urinary sodium excretion. Participants will also be invited to collect 24-hour urine 3 days in a row.
* To collect ons single fecal collection for the determination of the gut microbiota
* To participate in an intervention trial examining the effects of Vitamin K supplementation versus placebo on cardiovascular risk markers.

ELIGIBILITY:
Inclusion Criteria:

* Have participated in the Inter99 Baseline examination.

Exclusion Criteria:

* Physically or cognitively unable to participate in the 3-hour clinical follow-up study.

Ages: 50 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Former participants of the Inter99 cohort, now aged 50-80 years, will be re-invited to participate in the Inter99-20-year follow-up study. A search of the Danish nationwide civil register (CPR register) in December 2019 showed that 6,004 (88.5%) participants reside in Denmark are currently alive. Based on our experience, we expect that at least 4,000 incl. 500 or more T2D patients will participate in the follow-up study. All participants are invited to a follow-up health examination in CCRP located in Glostrup.
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2021-09-13 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular events (MACE) (Register data) | As data are collected from registers, the events are registered as they occur up until 1 Jan 2020.
  Composite endpoint of cardiovascular mortality, nonfatal myocardial infarction and nonfatal stroke (3 points MACE). Data are retrieved from the Danish national registers as described in the "study population" section.

SECONDARY OUTCOMES:
Type 2 diabetes incidence (register data) | As data are collected from registers, the events are registered as they occur up until 1 Jan 2020.
  Data are retrieved from the Danish national registers as described in the "study population" section.
Diabetic retinopathy (Optos) | Measured one time during the clinical follow-up study (Day 1).
  Assessed in each participant at the clinical follow-up
Liver stiffness (FibroScan) | Measured one time during the clinical follow-up study (Day 1).
  Assessed in each participant at the clinical follow-up
Heart rate variability (Vagus device) | Assessed in each participant at the clinical follow-up (Day 1).
  Assessed in each participant during the clinical follow-up study.
Pulse wave velocity (SphygmoCor) | Assessed in each participant at the clinical follow-up (Day 1).
  Assessed in each participant during the clinical follow-up study.
Hypertension (blood pressure) | Assessed in each participant at the clinical follow-up (Day 1).
  Assessed in each participant during the clinical follow-up study.
Physical function (sit to stand test) | Assessed in each participant at the clinical follow-up (Day 1).
  Assessed in each participant during the clinical follow-up study.
Handgrip strength (Handgrip dynamometer) | Assessed in each participant at the clinical follow-up (Day 1).
  Assessed in each participant during the clinical follow-up study.
Body composition using bioelectrical impedance technology (InBody770) | Assessed in each participant at the clinical follow-up (Day 1).
  Assessed in each participant during the clinical follow-up study.
Total daily physical energy expenditure (Sens Motion) | Assessed in each participant at the clinical follow-up (Day 1).
  Assessed in each participant that accepts to participate in the sub study with an activity monitor.
Glycemic variability (CGM) | Assessed in each participant at the clinical follow-up (Day 1).
  Assessed in each participant that accepts to participate in the sub study with a continuous glucose monitor.
Total daily energy intake (Diet registration) | Assessed in each participant at the clinical follow-up (Day 1).
  Assessed in each participant that accepts to participate in the sub study with the 24h diet registration.
Coronary artery calcification score (CT scan) | Assessed in each participant at the clinical follow-up (Day 1).
  Assessed in each participant that accepts to have their heart CT scanned. Total Coronary artery calcification (CAC) score (unit: Agatston score) in the coronary arteries, assessed by non-contrast Cardiac CT scans. A high score reflects high degree of calcification in the coronary arteries and increased risk of coronary artery disease.
Albumin excretion rate (urine samples) | Assessed in each participant at the clinical follow-up (Day 1).
  Assessed from urine samples drawn from each participant during the clinical follow-up study.
Chronic Kidney Disease (CKD) Stage 3/4/5 (Blood samples) | Assessed in each participant at the clinical follow-up (Day 1).
  Assessed from blood samples drawn from each participant during the clinical follow-up study.

CONTACTS AND LOCATIONS:
Overall Officials: Allan A Vaag, D.M.Sc/D.Sc, Principal Investigator — Steno Diabetes Center Copenhagen, The Capital Region of Denmark; Allan Linneberg, PhD, Study Chair — Center for Clinical Research and Prevention, The Capital Region of Denmark
Locations (1):
- Center for Klinisk Forskning og Forebyggelse, Glostrup Municipality, Denmark

REFERENCES:
- [Background] Gedebjerg A, Almdal TP, Berencsi K, Rungby J, Nielsen JS, Witte DR, Friborg S, Brandslund I, Vaag A, Beck-Nielsen H, Sorensen HT, Thomsen RW. Prevalence of micro- and macrovascular diabetes complications at time of type 2 diabetes diagnosis and associated clinical characteristics: A cross-sectional baseline study of 6958 patients in the Danish DD2 cohort. J Diabetes Complications. 2018 Jan;32(1):34-40. doi: 10.1016/j.jdiacomp.2017.09.010. Epub 2017 Sep 19. PMID 29107454
- [Background] Mahajan A, Taliun D, Thurner M, Robertson NR, Torres JM, Rayner NW, Payne AJ, Steinthorsdottir V, Scott RA, Grarup N, Cook JP, Schmidt EM, Wuttke M, Sarnowski C, Magi R, Nano J, Gieger C, Trompet S, Lecoeur C, Preuss MH, Prins BP, Guo X, Bielak LF, Below JE, Bowden DW, Chambers JC, Kim YJ, Ng MCY, Petty LE, Sim X, Zhang W, Bennett AJ, Bork-Jensen J, Brummett CM, Canouil M, Ec Kardt KU, Fischer K, Kardia SLR, Kronenberg F, Lall K, Liu CT, Locke AE, Luan J, Ntalla I, Nylander V, Schonherr S, Schurmann C, Yengo L, Bottinger EP, Brandslund I, Christensen C, Dedoussis G, Florez JC, Ford I, Franco OH, Frayling TM, Giedraitis V, Hackinger S, Hattersley AT, Herder C, Ikram MA, Ingelsson M, Jorgensen ME, Jorgensen T, Kriebel J, Kuusisto J, Ligthart S, Lindgren CM, Linneberg A, Lyssenko V, Mamakou V, Meitinger T, Mohlke KL, Morris AD, Nadkarni G, Pankow JS, Peters A, Sattar N, Stancakova A, Strauch K, Taylor KD, Thorand B, Thorleifsson G, Thorsteinsdottir U, Tuomilehto J, Witte DR, Dupuis J, Peyser PA, Zeggini E, Loos RJF, Froguel P, Ingelsson E, Lind L, Groop L, Laakso M, Collins FS, Jukema JW, Palmer CNA, Grallert H, Metspalu A, Dehghan A, Kottgen A, Abecasis GR, Meigs JB, Rotter JI, Marchini J, Pedersen O, Hansen T, Langenberg C, Wareham NJ, Stefansson K, Gloyn AL, Morris AP, Boehnke M, McCarthy MI. Fine-mapping type 2 diabetes loci to single-variant resolution using high-density imputation and islet-specific epigenome maps. Nat Genet. 2018 Nov;50(11):1505-1513. doi: 10.1038/s41588-018-0241-6. Epub 2018 Oct 8. PMID 30297969
- [Background] Wu L, Feng X, He A, Ding Y, Zhou X, Xu Z. Prenatal exposure to the Great Chinese Famine and mid-age hypertension. PLoS One. 2017 May 12;12(5):e0176413. doi: 10.1371/journal.pone.0176413. eCollection 2017. PMID 28498832
- [Background] Lumey LH, Khalangot MD, Vaiserman AM. Association between type 2 diabetes and prenatal exposure to the Ukraine famine of 1932-33: a retrospective cohort study. Lancet Diabetes Endocrinol. 2015 Oct;3(10):787-94. doi: 10.1016/S2213-8587(15)00279-X. Epub 2015 Sep 3. PMID 26342852
- [Background] Li Y, He Y, Qi L, Jaddoe VW, Feskens EJ, Yang X, Ma G, Hu FB. Exposure to the Chinese famine in early life and the risk of hyperglycemia and type 2 diabetes in adulthood. Diabetes. 2010 Oct;59(10):2400-6. doi: 10.2337/db10-0385. Epub 2010 Jul 9. PMID 20622161
- [Background] Ravelli AC, van der Meulen JH, Michels RP, Osmond C, Barker DJ, Hales CN, Bleker OP. Glucose tolerance in adults after prenatal exposure to famine. Lancet. 1998 Jan 17;351(9097):173-7. doi: 10.1016/s0140-6736(97)07244-9. PMID 9449872
- [Background] Tarry-Adkins JL, Ozanne SE. Nutrition in early life and age-associated diseases. Ageing Res Rev. 2017 Oct;39:96-105. doi: 10.1016/j.arr.2016.08.003. Epub 2016 Sep 1. PMID 27594376
- [Background] Ozanne SE, Constancia M. Mechanisms of disease: the developmental origins of disease and the role of the epigenotype. Nat Clin Pract Endocrinol Metab. 2007 Jul;3(7):539-46. doi: 10.1038/ncpendmet0531. PMID 17581623
- [Background] Dumortier O, Blondeau B, Duvillie B, Reusens B, Breant B, Remacle C. Different mechanisms operating during different critical time-windows reduce rat fetal beta cell mass due to a maternal low-protein or low-energy diet. Diabetologia. 2007 Dec;50(12):2495-503. doi: 10.1007/s00125-007-0811-0. Epub 2007 Sep 19. PMID 17882398
- [Background] Ndiaye FK, Ortalli A, Canouil M, Huyvaert M, Salazar-Cardozo C, Lecoeur C, Verbanck M, Pawlowski V, Boutry R, Durand E, Rabearivelo I, Sand O, Marselli L, Kerr-Conte J, Chandra V, Scharfmann R, Poulain-Godefroy O, Marchetti P, Pattou F, Abderrahmani A, Froguel P, Bonnefond A. Expression and functional assessment of candidate type 2 diabetes susceptibility genes identify four new genes contributing to human insulin secretion. Mol Metab. 2017 Apr 8;6(6):459-470. doi: 10.1016/j.molmet.2017.03.011. eCollection 2017 Jun. PMID 28580277
- [Background] Warrington NM, Beaumont RN, Horikoshi M, Day FR, Helgeland O, Laurin C, Bacelis J, Peng S, Hao K, Feenstra B, Wood AR, Mahajan A, Tyrrell J, Robertson NR, Rayner NW, Qiao Z, Moen GH, Vaudel M, Marsit CJ, Chen J, Nodzenski M, Schnurr TM, Zafarmand MH, Bradfield JP, Grarup N, Kooijman MN, Li-Gao R, Geller F, Ahluwalia TS, Paternoster L, Rueedi R, Huikari V, Hottenga JJ, Lyytikainen LP, Cavadino A, Metrustry S, Cousminer DL, Wu Y, Thiering E, Wang CA, Have CT, Vilor-Tejedor N, Joshi PK, Painter JN, Ntalla I, Myhre R, Pitkanen N, van Leeuwen EM, Joro R, Lagou V, Richmond RC, Espinosa A, Barton SJ, Inskip HM, Holloway JW, Santa-Marina L, Estivill X, Ang W, Marsh JA, Reichetzeder C, Marullo L, Hocher B, Lunetta KL, Murabito JM, Relton CL, Kogevinas M, Chatzi L, Allard C, Bouchard L, Hivert MF, Zhang G, Muglia LJ, Heikkinen J; EGG Consortium; Morgen CS, van Kampen AHC, van Schaik BDC, Mentch FD, Langenberg C, Luan J, Scott RA, Zhao JH, Hemani G, Ring SM, Bennett AJ, Gaulton KJ, Fernandez-Tajes J, van Zuydam NR, Medina-Gomez C, de Haan HG, Rosendaal FR, Kutalik Z, Marques-Vidal P, Das S, Willemsen G, Mbarek H, Muller-Nurasyid M, Standl M, Appel EVR, Fonvig CE, Trier C, van Beijsterveldt CEM, Murcia M, Bustamante M, Bonas-Guarch S, Hougaard DM, Mercader JM, Linneberg A, Schraut KE, Lind PA, Medland SE, Shields BM, Knight BA, Chai JF, Panoutsopoulou K, Bartels M, Sanchez F, Stokholm J, Torrents D, Vinding RK, Willems SM, Atalay M, Chawes BL, Kovacs P, Prokopenko I, Tuke MA, Yaghootkar H, Ruth KS, Jones SE, Loh PR, Murray A, Weedon MN, Tonjes A, Stumvoll M, Michaelsen KF, Eloranta AM, Lakka TA, van Duijn CM, Kiess W, Korner A, Niinikoski H, Pahkala K, Raitakari OT, Jacobsson B, Zeggini E, Dedoussis GV, Teo YY, Saw SM, Montgomery GW, Campbell H, Wilson JF, Vrijkotte TGM, Vrijheid M, de Geus EJCN, Hayes MG, Kadarmideen HN, Holm JC, Beilin LJ, Pennell CE, Heinrich J, Adair LS, Borja JB, Mohlke KL, Eriksson JG, Widen EE, Hattersley AT, Spector TD, Kahonen M, Viikari JS, Lehtimaki T, Boomsma DI, Sebert S, Vollenweider P, Sorensen TIA, Bisgaard H, Bonnelykke K, Murray JC, Melbye M, Nohr EA, Mook-Kanamori DO, Rivadeneira F, Hofman A, Felix JF, Jaddoe VWV, Hansen T, Pisinger C, Vaag AA, Pedersen O, Uitterlinden AG, Jarvelin MR, Power C, Hypponen E, Scholtens DM, Lowe WL Jr, Davey Smith G, Timpson NJ, Morris AP, Wareham NJ, Hakonarson H, Grant SFA, Frayling TM, Lawlor DA, Njolstad PR, Johansson S, Ong KK, McCarthy MI, Perry JRB, Evans DM, Freathy RM. Maternal and fetal genetic effects on birth weight and their relevance to cardio-metabolic risk factors. Nat Genet. 2019 May;51(5):804-814. doi: 10.1038/s41588-019-0403-1. Epub 2019 May 1. PMID 31043758
- [Background] Barker DJ, Martyn CN, Osmond C, Hales CN, Fall CH. Growth in utero and serum cholesterol concentrations in adult life. BMJ. 1993 Dec 11;307(6918):1524-7. doi: 10.1136/bmj.307.6918.1524. PMID 8274921
- [Background] Painter RC, de Rooij SR, Bossuyt PM, Simmers TA, Osmond C, Barker DJ, Bleker OP, Roseboom TJ. Early onset of coronary artery disease after prenatal exposure to the Dutch famine. Am J Clin Nutr. 2006 Aug;84(2):322-7; quiz 466-7. doi: 10.1093/ajcn/84.1.322. PMID 16895878
- [Background] Tamashiro KL, Terrillion CE, Hyun J, Koenig JI, Moran TH. Prenatal stress or high-fat diet increases susceptibility to diet-induced obesity in rat offspring. Diabetes. 2009 May;58(5):1116-25. doi: 10.2337/db08-1129. Epub 2009 Feb 2. PMID 19188431
- [Background] Berge LN, Arnesen E, Forsdahl A. Pregnancy related changes in some cardiovascular risk factors. Acta Obstet Gynecol Scand. 1996 May;75(5):439-42. doi: 10.3109/00016349609033350. PMID 8677767
- [Background] Osmond C, Barker DJ, Winter PD, Fall CH, Simmonds SJ. Early growth and death from cardiovascular disease in women. BMJ. 1993 Dec 11;307(6918):1519-24. doi: 10.1136/bmj.307.6918.1519. PMID 8274920
- [Background] Leibson CL, Burke JP, Ransom JE, Forsgren J, Melton J 3rd, Bailey KR, Palumbo PJ. Relative risk of mortality associated with diabetes as a function of birth weight. Diabetes Care. 2005 Dec;28(12):2839-43. doi: 10.2337/diacare.28.12.2839. PMID 16306542
- [Background] Hellstrom A, Hard AL, Niklasson A, Svensson E, Jacobsson B. Abnormal retinal vascularisation in preterm children as a general vascular phenomenon. Lancet. 1998 Dec 5;352(9143):1827. doi: 10.1016/S0140-6736(05)79889-5. No abstract available. PMID 9851388
- [Background] Liew G, Wang JJ, Duncan BB, Klein R, Sharrett AR, Brancati F, Yeh HC, Mitchell P, Wong TY; Atherosclerosis Risk in Communities Study. Low birthweight is associated with narrower arterioles in adults. Hypertension. 2008 Apr;51(4):933-8. doi: 10.1161/HYPERTENSIONAHA.107.101584. Epub 2008 Feb 11. PMID 18268137
- [Background] Fedotkina O, Luk A, Jain R, Prasad RB, Shungin D, Simo-Servat O, Ozgumus T, Cherviakova L, Khalimon N, Svietleisha T, Buldenko T, Kravchenko V, Hernandez C, Jain D, Simo R, Artner I, Nilsson PM, Khalangot MD, Vaiserman AM, Chan J, Vaag A, Lyssenko V. Perinatal famine is associated with excess risk of proliferative retinopathy in patients with type 2 diabetes. Acta Ophthalmol. 2022 Mar;100(2):e539-e545. doi: 10.1111/aos.14948. Epub 2021 Jun 24. PMID 34169655
- [Background] Eriksson JG, Salonen MK, Kajantie E, Osmond C. Prenatal Growth and CKD in Older Adults: Longitudinal Findings From the Helsinki Birth Cohort Study, 1924-1944. Am J Kidney Dis. 2018 Jan;71(1):20-26. doi: 10.1053/j.ajkd.2017.06.030. Epub 2017 Aug 23. PMID 28838764
- [Background] Souza LV, Oliveira V, De Meneck F, Grotti Clemente AP, Strufaldi MW, Franco MD. Birth Weight and Its Relationship with the Cardiac Autonomic Balance in Healthy Children. PLoS One. 2017 Jan 17;12(1):e0167328. doi: 10.1371/journal.pone.0167328. eCollection 2017. PMID 28095501
- [Background] Younossi Z, Anstee QM, Marietti M, Hardy T, Henry L, Eslam M, George J, Bugianesi E. Global burden of NAFLD and NASH: trends, predictions, risk factors and prevention. Nat Rev Gastroenterol Hepatol. 2018 Jan;15(1):11-20. doi: 10.1038/nrgastro.2017.109. Epub 2017 Sep 20. PMID 28930295
- [Background] Younossi ZM, Koenig AB, Abdelatif D, Fazel Y, Henry L, Wymer M. Global epidemiology of nonalcoholic fatty liver disease-Meta-analytic assessment of prevalence, incidence, and outcomes. Hepatology. 2016 Jul;64(1):73-84. doi: 10.1002/hep.28431. Epub 2016 Feb 22. PMID 26707365
- [Background] Lauridsen BK, Stender S, Kristensen TS, Kofoed KF, Kober L, Nordestgaard BG, Tybjaerg-Hansen A. Liver fat content, non-alcoholic fatty liver disease, and ischaemic heart disease: Mendelian randomization and meta-analysis of 279 013 individuals. Eur Heart J. 2018 Feb 1;39(5):385-393. doi: 10.1093/eurheartj/ehx662. PMID 29228164
- [Background] Mikalsen IB, Halvorsen T, Juliusson PB, Magnus M, Nystad W, Stensrud T, Stordal K, Vollsaeter M, Oymar K. Early life growth and associations with lung function and bronchial hyperresponsiveness at 11-years of age. Respir Med. 2021 Feb;177:106305. doi: 10.1016/j.rmed.2021.106305. Epub 2021 Jan 8. PMID 33482491
- [Background] Vujkovic M, Keaton JM, Lynch JA, Miller DR, Zhou J, Tcheandjieu C, Huffman JE, Assimes TL, Lorenz K, Zhu X, Hilliard AT, Judy RL, Huang J, Lee KM, Klarin D, Pyarajan S, Danesh J, Melander O, Rasheed A, Mallick NH, Hameed S, Qureshi IH, Afzal MN, Malik U, Jalal A, Abbas S, Sheng X, Gao L, Kaestner KH, Susztak K, Sun YV, DuVall SL, Cho K, Lee JS, Gaziano JM, Phillips LS, Meigs JB, Reaven PD, Wilson PW, Edwards TL, Rader DJ, Damrauer SM, O'Donnell CJ, Tsao PS; HPAP Consortium; Regeneron Genetics Center; VA Million Veteran Program; Chang KM, Voight BF, Saleheen D. Discovery of 318 new risk loci for type 2 diabetes and related vascular outcomes among 1.4 million participants in a multi-ancestry meta-analysis. Nat Genet. 2020 Jul;52(7):680-691. doi: 10.1038/s41588-020-0637-y. Epub 2020 Jun 15. PMID 32541925
- [Background] Horikoshi M, Yaghootkar H, Mook-Kanamori DO, Sovio U, Taal HR, Hennig BJ, Bradfield JP, St Pourcain B, Evans DM, Charoen P, Kaakinen M, Cousminer DL, Lehtimaki T, Kreiner-Moller E, Warrington NM, Bustamante M, Feenstra B, Berry DJ, Thiering E, Pfab T, Barton SJ, Shields BM, Kerkhof M, van Leeuwen EM, Fulford AJ, Kutalik Z, Zhao JH, den Hoed M, Mahajan A, Lindi V, Goh LK, Hottenga JJ, Wu Y, Raitakari OT, Harder MN, Meirhaeghe A, Ntalla I, Salem RM, Jameson KA, Zhou K, Monies DM, Lagou V, Kirin M, Heikkinen J, Adair LS, Alkuraya FS, Al-Odaib A, Amouyel P, Andersson EA, Bennett AJ, Blakemore AI, Buxton JL, Dallongeville J, Das S, de Geus EJ, Estivill X, Flexeder C, Froguel P, Geller F, Godfrey KM, Gottrand F, Groves CJ, Hansen T, Hirschhorn JN, Hofman A, Hollegaard MV, Hougaard DM, Hypponen E, Inskip HM, Isaacs A, Jorgensen T, Kanaka-Gantenbein C, Kemp JP, Kiess W, Kilpelainen TO, Klopp N, Knight BA, Kuzawa CW, McMahon G, Newnham JP, Niinikoski H, Oostra BA, Pedersen L, Postma DS, Ring SM, Rivadeneira F, Robertson NR, Sebert S, Simell O, Slowinski T, Tiesler CM, Tonjes A, Vaag A, Viikari JS, Vink JM, Vissing NH, Wareham NJ, Willemsen G, Witte DR, Zhang H, Zhao J; Meta-Analyses of Glucose- and Insulin-related traits Consortium (MAGIC); Wilson JF, Stumvoll M, Prentice AM, Meyer BF, Pearson ER, Boreham CA, Cooper C, Gillman MW, Dedoussis GV, Moreno LA, Pedersen O, Saarinen M, Mohlke KL, Boomsma DI, Saw SM, Lakka TA, Korner A, Loos RJ, Ong KK, Vollenweider P, van Duijn CM, Koppelman GH, Hattersley AT, Holloway JW, Hocher B, Heinrich J, Power C, Melbye M, Guxens M, Pennell CE, Bonnelykke K, Bisgaard H, Eriksson JG, Widen E, Hakonarson H, Uitterlinden AG, Pouta A, Lawlor DA, Smith GD, Frayling TM, McCarthy MI, Grant SF, Jaddoe VW, Jarvelin MR, Timpson NJ, Prokopenko I, Freathy RM; Early Growth Genetics (EGG) Consortium. New loci associated with birth weight identify genetic links between intrauterine growth and adult height and metabolism. Nat Genet. 2013 Jan;45(1):76-82. doi: 10.1038/ng.2477. Epub 2012 Dec 2. PMID 23202124
- [Background] Horikoshi M, Beaumont RN, Day FR, Warrington NM, Kooijman MN, Fernandez-Tajes J, Feenstra B, van Zuydam NR, Gaulton KJ, Grarup N, Bradfield JP, Strachan DP, Li-Gao R, Ahluwalia TS, Kreiner E, Rueedi R, Lyytikainen LP, Cousminer DL, Wu Y, Thiering E, Wang CA, Have CT, Hottenga JJ, Vilor-Tejedor N, Joshi PK, Boh ETH, Ntalla I, Pitkanen N, Mahajan A, van Leeuwen EM, Joro R, Lagou V, Nodzenski M, Diver LA, Zondervan KT, Bustamante M, Marques-Vidal P, Mercader JM, Bennett AJ, Rahmioglu N, Nyholt DR, Ma RCW, Tam CHT, Tam WH; CHARGE Consortium Hematology Working Group; Ganesh SK, van Rooij FJ, Jones SE, Loh PR, Ruth KS, Tuke MA, Tyrrell J, Wood AR, Yaghootkar H, Scholtens DM, Paternoster L, Prokopenko I, Kovacs P, Atalay M, Willems SM, Panoutsopoulou K, Wang X, Carstensen L, Geller F, Schraut KE, Murcia M, van Beijsterveldt CE, Willemsen G, Appel EVR, Fonvig CE, Trier C, Tiesler CM, Standl M, Kutalik Z, Bonas-Guarch S, Hougaard DM, Sanchez F, Torrents D, Waage J, Hollegaard MV, de Haan HG, Rosendaal FR, Medina-Gomez C, Ring SM, Hemani G, McMahon G, Robertson NR, Groves CJ, Langenberg C, Luan J, Scott RA, Zhao JH, Mentch FD, MacKenzie SM, Reynolds RM; Early Growth Genetics (EGG) Consortium; Lowe WL Jr, Tonjes A, Stumvoll M, Lindi V, Lakka TA, van Duijn CM, Kiess W, Korner A, Sorensen TI, Niinikoski H, Pahkala K, Raitakari OT, Zeggini E, Dedoussis GV, Teo YY, Saw SM, Melbye M, Campbell H, Wilson JF, Vrijheid M, de Geus EJ, Boomsma DI, Kadarmideen HN, Holm JC, Hansen T, Sebert S, Hattersley AT, Beilin LJ, Newnham JP, Pennell CE, Heinrich J, Adair LS, Borja JB, Mohlke KL, Eriksson JG, Widen EE, Kahonen M, Viikari JS, Lehtimaki T, Vollenweider P, Bonnelykke K, Bisgaard H, Mook-Kanamori DO, Hofman A, Rivadeneira F, Uitterlinden AG, Pisinger C, Pedersen O, Power C, Hypponen E, Wareham NJ, Hakonarson H, Davies E, Walker BR, Jaddoe VW, Jarvelin MR, Grant SF, Vaag AA, Lawlor DA, Frayling TM, Davey Smith G, Morris AP, Ong KK, Felix JF, Timpson NJ, Perry JR, Evans DM, McCarthy MI, Freathy RM. Genome-wide associations for birth weight and correlations with adult disease. Nature. 2016 Oct 13;538(7624):248-252. doi: 10.1038/nature19806. Epub 2016 Sep 28. PMID 27680694
- [Background] Carstensen B, Ronn PF, Jorgensen ME. Prevalence, incidence and mortality of type 1 and type 2 diabetes in Denmark 1996-2016. BMJ Open Diabetes Res Care. 2020 May;8(1):e001071. doi: 10.1136/bmjdrc-2019-001071. PMID 32475839
- [Background] Grann AF, Erichsen R, Nielsen AG, Froslev T, Thomsen RW. Existing data sources for clinical epidemiology: The clinical laboratory information system (LABKA) research database at Aarhus University, Denmark. Clin Epidemiol. 2011 Apr 1;3:133-8. doi: 10.2147/CLEP.S17901. PMID 21487452
- [Background] Andersen TF, Madsen M, Jorgensen J, Mellemkjoer L, Olsen JH. The Danish National Hospital Register. A valuable source of data for modern health sciences. Dan Med Bull. 1999 Jun;46(3):263-8. PMID 10421985
- [Background] Ahlqvist E, Storm P, Karajamaki A, Martinell M, Dorkhan M, Carlsson A, Vikman P, Prasad RB, Aly DM, Almgren P, Wessman Y, Shaat N, Spegel P, Mulder H, Lindholm E, Melander O, Hansson O, Malmqvist U, Lernmark A, Lahti K, Forsen T, Tuomi T, Rosengren AH, Groop L. Novel subgroups of adult-onset diabetes and their association with outcomes: a data-driven cluster analysis of six variables. Lancet Diabetes Endocrinol. 2018 May;6(5):361-369. doi: 10.1016/S2213-8587(18)30051-2. Epub 2018 Mar 5. PMID 29503172
- [Background] Faerch K, Witte DR, Tabak AG, Perreault L, Herder C, Brunner EJ, Kivimaki M, Vistisen D. Trajectories of cardiometabolic risk factors before diagnosis of three subtypes of type 2 diabetes: a post-hoc analysis of the longitudinal Whitehall II cohort study. Lancet Diabetes Endocrinol. 2013 Sep;1(1):43-51. doi: 10.1016/S2213-8587(13)70008-1. Epub 2013 Feb 21. PMID 24622266
- [Result] Vaag AA, Grunnet LG, Arora GP, Brons C. The thrifty phenotype hypothesis revisited. Diabetologia. 2012 Aug;55(8):2085-8. doi: 10.1007/s00125-012-2589-y. Epub 2012 May 30. PMID 22643933
- [Result] Jorgensen T, Borch-Johnsen K, Thomsen TF, Ibsen H, Glumer C, Pisinger C. A randomized non-pharmacological intervention study for prevention of ischaemic heart disease: baseline results Inter99. Eur J Cardiovasc Prev Rehabil. 2003 Oct;10(5):377-86. doi: 10.1097/01.hjr.0000096541.30533.82. PMID 14663300
- [Result] Lau C, Vistisen D, Toft U, Tetens I, Glumer C, Pedersen O, Jorgensen T, Borch-Johnsen K. The effects of adding group-based lifestyle counselling to individual counselling on changes in plasma glucose levels in a randomized controlled trial: the Inter99 study. Diabetes Metab. 2011 Dec;37(6):546-52. doi: 10.1016/j.diabet.2011.06.001. Epub 2011 Sep 6. PMID 21900030
- [Result] Lau CJ, Pisinger C, Husemoen LLN, Jacobsen RK, Linneberg A, Jorgensen T, Glumer C. Effect of general health screening and lifestyle counselling on incidence of diabetes in general population: Inter99 randomised trial. Prev Med. 2016 Oct;91:172-179. doi: 10.1016/j.ypmed.2016.08.016. Epub 2016 Aug 8. PMID 27514243
- [Result] Jorgensen T, Jacobsen RK, Toft U, Aadahl M, Glumer C, Pisinger C. Effect of screening and lifestyle counselling on incidence of ischaemic heart disease in general population: Inter99 randomised trial. BMJ. 2014 Jun 9;348:g3617. doi: 10.1136/bmj.g3617. PMID 24912589
- [Result] Pilgaard K, Faerch K, Poulsen P, Larsen C, Andersson EA, Pisinger C, Toft U, Aadahl M, Pedersen O, Hansen T, Borch-Johnsen K, Vaag A, Jorgensen T. Impact of size at birth and prematurity on adult anthropometry in 4744 middle-aged Danes - The Inter99 study. J Dev Orig Health Dis. 2010 Oct;1(5):319-28. doi: 10.1017/S2040174410000413. PMID 25141935
- [Result] Pilgaard K, Faerch K, Carstensen B, Poulsen P, Pisinger C, Pedersen O, Witte DR, Hansen T, Jorgensen T, Vaag A. Low birthweight and premature birth are both associated with type 2 diabetes in a random sample of middle-aged Danes. Diabetologia. 2010 Dec;53(12):2526-30. doi: 10.1007/s00125-010-1917-3. Epub 2010 Sep 22. PMID 20859612
- [Result] Munch IC, Larsen M, Kessel L, Borch-Johnsen K, Lund-Andersen H, Glumer C. Cumulative glycemia and microangiopathy in subjects with impaired glucose regulation in the Inter99 study. Diabetes Res Clin Pract. 2011 Feb;91(2):226-32. doi: 10.1016/j.diabres.2010.10.017. Epub 2010 Dec 3. PMID 21130512
- [Result] Engberg S, Vistisen D, Lau C, Glumer C, Jorgensen T, Pedersen O, Borch-Johnsen K. Progression to impaired glucose regulation and diabetes in the population-based Inter99 study. Diabetes Care. 2009 Apr;32(4):606-11. doi: 10.2337/dc08-1869. Epub 2008 Dec 29. PMID 19114617
- [Derived] Bjornsbo KS, Brons C, Aadahl M, Kampmann FB, Friis Bryde Nielsen C, Lundbergh B, Wibaek R, Karhus LL, Madsen AL, Hansen CS, Norgaard K, Jorgensen NR, Suetta C, Kjaer M, Grarup N, Kanters J, Larsen M, Kober L, Kofoed KF, Loos R, Hansen T, Linneberg A, Vaag A. Protocol for the combined cardiometabolic deep phenotyping and registry-based 20-year follow-up study of the Inter99 cohort. BMJ Open. 2024 Jan 29;14(1):e078501. doi: 10.1136/bmjopen-2023-078501. PMID 38286704